CLINICAL TRIAL: NCT02390531
Title: Phase 1 Trial of Bevacizumab Treatment for Severe Retinopathy of Prematurity
Acronym: ROP1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Pediatric Eye Disease Investigator Group (Network); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ROP1; 2U10EY011751 (NIH)
Record Dates: First submitted 2015-02-17; First posted 2015-03-17 (Estimated); Results first posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Retinopathy of Prematurity
Keywords: Retinopathy of Prematurity; Bevacizumab; ROP
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Bevacizumab

STUDY DESIGN:
Intervention Model Description: 8 bevacizumab doses were evaluated in this dose de-escalation study in the following dosage amounts: 0.250mg, 0.125mg, 0.063mg, 0.031mg, 0.016mg, 0.008mg, 0.004mg, 0.002mg. Each dose was planned to be used in up to 14 infants to ensure at least 10 infants with 4-week outcomes
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Bevacizumab 0.250 mg (Experimental): Dosage of injected Bevacizumab to be studied
  Interventions: Drug: Bevacizumab
- Bevacizumab 0.125 mg (Experimental): Dosage of injected Bevacizumab to be studied
  Interventions: Drug: Bevacizumab
- Bevacizumab 0.063 mg (Experimental): Dosage of injected Bevacizumab to be studied
  Interventions: Drug: Bevacizumab
- Bevacizumab 0.031 mg (Experimental): Dosage of injected Bevacizumab to be studied
  Interventions: Drug: Bevacizumab
- Bevacizumab 0.016 mg (Experimental): Dosage of injected Bevacizumab to be studied
  Interventions: Drug: Bevacizumab
- Bevacizumab 0.008 mg (Experimental): Dosage of injected Bevacizumab to be studied
  Interventions: Drug: Bevacizumab
- Bevacizumab 0.004 mg (Experimental): Dosage of injected Bevacizumab to be studied
  Interventions: Drug: Bevacizumab
- Bevacizumab 0.002 mg (Experimental): Dosage of injected Bevacizumab to be studied
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Varying dosages in 10µl
  Other Names: Avastin

SUMMARY:
The purpose of this study is to find a dose of intravitreal bevacizumab that is lower than currently used for severe retinopathy of prematurity (ROP), is effective in this study, and can be tested in future larger studies.

DETAILED DESCRIPTION:
Despite promising initial results using empirical doses of bevacizumab based on half the adult dose for treatment of acute severe ROP, little is known about lower doses of bevacizumab for ROP. An increasing number of ophthalmologists are treating premature infants with severe ROP using bevacizumab. Given the potential systemic and ocular adverse effects of intravitreal bevacizumab injections, determining a lower effective dose of bevacizumab is an important next step. The proposed study will test progressively lower doses to find a dose to take forward to a future larger study.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 ROP; defined as:

   * Zone I, any stage ROP with plus disease, or
   * Zone I, stage 3 ROP without plus disease, or
   * Zone II, stage 2 or 3 ROP with plus disease
2. No previous treatment for ROP in the study eye; no previous bevacizumab treatment in the non-study eye

Exclusion Criteria:

The following exclusions apply to the study eye:

1. Nasolacrimal duct obstruction
2. Major ocular anomalies (e.g., cataract, coloboma)
3. Any opacity that precludes an adequate view of the retina

If purulent ocular discharge is present in either eye, then the infant is ineligible.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2021-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David K Wallace, MD, MPH, Study Chair — Indiana University
Locations (11):
- United States (11):
  - The Emory Eye Center, Atlanta, Georgia
  - Riley Hospital for Children, Indianapolis, Indiana
  - Wilmer Institute, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Duke University Eye Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Pediatric Ophthalmology Associates, Inc., Columbus, Ohio
  - Dean A. McGee Eye Institute, University of Oklahoma, Oklahoma City, Oklahoma
  - Texas Children's Hospital - Dept. Of Ophthalmology, Houston, Texas
  - University of Utah Moran Eye Center, Salt Lake City, Utah
  - Virginia Pediatric Eye Center, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH data sharing policy, a de-identified database is placed in the public domain on the PEDIG public website after the completion of each protocol and publication of the primary manuscript.
Time Frame: Data will be made available after publication of each primary manuscript.
Access Criteria: Users accessing the data must enter an email address.

REFERENCES:
- [Background] Wallace DK, Kraker RT, Freedman SF, Crouch ER, Hutchinson AK, Bhatt AR, Rogers DL, Yang MB, Haider KM, VanderVeen DK, Siatkowski RM, Dean TW, Beck RW, Repka MX, Smith LE, Good WV, Hartnett ME, Kong L, Holmes JM; Pediatric Eye Disease Investigator Group (PEDIG). Assessment of Lower Doses of Intravitreous Bevacizumab for Retinopathy of Prematurity: A Phase 1 Dosing Study. JAMA Ophthalmol. 2017 Jun 1;135(6):654-656. doi: 10.1001/jamaophthalmol.2017.1055. PMID 28448664
- [Background] Kraker RT, Wallace DK, Beck RW, Saunders CT, Lorenzi E, Melia BM, Li Z; Pediatric Eye Disease Investigator Group. Choice of Dose Level for a Randomized Clinical Trial of Low-Dose Bevacizumab vs Laser for Type 1 Retinopathy of Prematurity. JAMA Ophthalmol. 2021 Oct 1;139(10):1143-1144. doi: 10.1001/jamaophthalmol.2021.3192. PMID 34410311
- [Result] Wallace DK, Dean TW, Hartnett ME, Kong L, Smith LE, Hubbard GB, McGregor ML, Jordan CO, Mantagos IS, Bell EF, Kraker RT; Pediatric Eye Disease Investigator Group. A Dosing Study of Bevacizumab for Retinopathy of Prematurity: Late Recurrences and Additional Treatments. Ophthalmology. 2018 Dec;125(12):1961-1966. doi: 10.1016/j.ophtha.2018.05.001. Epub 2018 Jun 7. PMID 29887334
- [Result] Crouch ER, Kraker RT, Wallace DK, Holmes JM, Repka MX, Collinge JE, Bremer DL, Gray ME, Smith HA, Steinkuller PG; Writing Committee for Pediatric Eye Disease Investigator Group. Secondary 12-Month Ocular Outcomes of a Phase 1 Dosing Study of Bevacizumab for Retinopathy of Prematurity. JAMA Ophthalmol. 2020 Jan 1;138(1):14-20. doi: 10.1001/jamaophthalmol.2019.4488. PMID 31697304
- [Result] Wallace DK, Kraker RT, Freedman SF, Crouch ER, Bhatt AR, Hartnett ME, Yang MB, Rogers DL, Hutchinson AK, VanderVeen DK, Haider KM, Siatkowski RM, Dean TW, Beck RW, Repka MX, Smith LE, Good WV, Kong L, Cotter SA, Holmes JM; Pediatric Eye Disease Investigator Group (PEDIG). Short-term Outcomes After Very Low-Dose Intravitreous Bevacizumab for Retinopathy of Prematurity. JAMA Ophthalmol. 2020 Jun 1;138(6):698-701. doi: 10.1001/jamaophthalmol.2020.0334. PMID 32324197
- See also: PEDIG Public Website — http://www.pedig.net

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Original reported enrollment was 121, however upon further review 2 patient identifiers were found to be the same patient, incorrectly enrolled twice, bringing the correct count to 120.
Groups:
- Bevacizumab (0.250 mg); Bevacizumab (0.125 mg); Bevacizumab (0.063 mg); Bevacizumab (0.031 mg); Bevacizumab (0.016 mg); Bevacizumab (0.008 mg); Bevacizumab (0.004 mg); Bevacizumab (0.002 mg): Dosage of injected Bevacizumab injected into study eye. When both eyes were treated, the fellow eye received the next higher dose than received by the study eye. More study eyes than fellow eyes were treated because some infants had type 1 ROP in one eye only.
Period: Overall Study
Arm/Group | Bevacizumab (0.250 mg) | Bevacizumab (0.125 mg) | Bevacizumab (0.063 mg) | Bevacizumab (0.031 mg) | Bevacizumab (0.016 mg) | Bevacizumab (0.008 mg) | Bevacizumab (0.004 mg) | Bevacizumab (0.002 mg)
Started | 11 | 16 | 24 | 10 | 14 | 9 | 12 | 24
Completed | 11 | 14 | 24 | 9 | 13 | 9 | 10 | 23
Not Completed | 0 | 2 | 0 | 1 | 1 | 0 | 2 | 1
Not completed — Death | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Bevacizumab (0.25 mg); Bevacizumab (0.125 mg); Bevacizumab (0.0625 mg); Bevacizumab (0.031 mg); Bevacizumab (0.016 mg); Bevacizumab (0.008 mg); Bevacizumab (0.004 mg); Bevacizumab (0.002 mg): Dosage of injected Bevacizumab to be studied
- Total: Total of all reporting groups
Arm/Group | Bevacizumab (0.25 mg) | Bevacizumab (0.125 mg) | Bevacizumab (0.0625 mg) | Bevacizumab (0.031 mg) | Bevacizumab (0.016 mg) | Bevacizumab (0.008 mg) | Bevacizumab (0.004 mg) | Bevacizumab (0.002 mg) | Total
Number analyzed (Participants) | 11 | 16 | 24 | 10 | 14 | 9 | 12 | 24 | 120
Age, Continuous [Mean (Standard Deviation); unit: Weeks] — Gestational Age in Weeks
  Weeks
    Gestational age at enrollment | 24.81 (1.49) | 25.21 (2.22) | 24.82 (1.42) | 24.73 (1.12) | 24.48 (1.14) | 24.63 (1.48) | 24.45 (1.23) | 25.14 (2.02) | 24.84 (1.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 12 | 4 | 3 | 7 | 3 | 10 | 49
  Male | 5 | 12 | 12 | 6 | 11 | 2 | 9 | 14 | 71
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7 | 10 | 12 | 2 | 9 | 3 | 7 | 15 | 65
  Black/African American | 2 | 2 | 3 | 4 | 2 | 2 | 2 | 2 | 19
  Hispanic or Latino | 2 | 3 | 3 | 2 | 2 | 1 | 2 | 2 | 17
  Asian | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 5
  Native Hawaiian/Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  American Indian/Alaskan Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  More than 1 race | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 4
  Unknown/Not Reported | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 3 | 7
Birth Weight [Mean (Standard Deviation); unit: grams] | 726.27 (219.23) | 801.31 (514.35) | 652.08 (156.88) | 680.60 (167.17) | 677.93 (147.02) | 539.44 (133.19) | 624.67 (155.14) | 722.00 (357.65) | 686.97 (281.43)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Treatment of ROP
Description: Success is defined as improvement* by the 4-day exam and no recurrence of type 1 ROP or severe neovascularization requiring additional treatment within 4 weeks of injection.
  * For infants with plus disease, improvement by the 4-day post-injection exam is defined as plus disease no longer being present. For infants with type 1 ROP without plus disease (i.e., zone I, stage 3), improvement by the 4-day post-injection exam is defined as: (1) a significant reduction in severity and/or extent of extraretinal neovascularization, and, (2) if pre-plus was present pre-injection, reduction in the degree of abnormal vascular dilation and/or tortuosity.
  A dose will be considered effective if it successfully treats at least 80% of subjects.
Time Frame: 4 weeks post-injection
Population: Seven infants were excluded (4 infants died prior to 4-week outcome examination; 1 failed, but it was not confirmed by second examiner; 1 was injected with the wrong dose in the study eye; and 1 had the fellow eye treated in the absence of type 1 ROP within one week of the study eye).
Measure: Count of Participants; unit: Participants
Groups:
- Bevacizumab: Dosage if injected Bevacizumab to be studied
  Bevacizumab: Varying dosages in 10µl
Arm/Group | Bevacizumab
Number analyzed (Participants) | 113
Participants
  0.250 mg Bevacizumab: number analyzed (Participants) | 11
  0.250 mg Bevacizumab | 11
  0.125 mg Bevacizumab: number analyzed (Participants) | 14
  0.125 mg Bevacizumab | 14
  0.063 mg Bevacizumab: number analyzed (Participants) | 24
  0.063 mg Bevacizumab | 21
  0.031 mg Bevacizumab: number analyzed (Participants) | 9
  0.031 mg Bevacizumab | 9
  0.016 mg Bevacizumab: number analyzed (Participants) | 13
  0.016 mg Bevacizumab | 13
  0.008 mg Bevacizumab: number analyzed (Participants) | 9
  0.008 mg Bevacizumab | 9
  0.004 mg Bevacizumab: number analyzed (Participants) | 10
  0.004 mg Bevacizumab | 9
  0.002 mg Bevacizumab: number analyzed (Participants) | 23
  0.002 mg Bevacizumab | 17

2. Secondary Outcome: Distribution of VEGF Levels
Description: The parents of each infant enrolled in the study will be given the option to participate in a study to measure levels of vascular endothelial growth factor (VEGF) and Avastin in the plasma. Participants in this optional study will have blood collected for analysis The distribution of VEGF and Avastin levels (median, range, and quartiles) will be described before injection, and at 2 weeks and 4 weeks post-injection. For each dosage level, at 2, and 4-weeks post-injection, the change from pre-injection will be calculated.
Time Frame: 2 weeks post-injection
Population: In this optional portion of the study, data is available for 66 infants.
Measure: Count of Participants; unit: Participants
Groups:
- Bevacizumab (0.0125 mg); Bevacizumab (0.0625 mg); Bevacizumab (0.031 mg); Bevacizumab (0.016 mg); Bevacizumab (0.008 mg); Bevacizumab (0.004 mg); Bevacizumab (0.002 mg): Dosage of injected Bevacizumab to be studied
Arm/Group | Bevacizumab (0.25 mg) | Bevacizumab (0.0125 mg) | Bevacizumab (0.0625 mg) | Bevacizumab (0.031 mg) | Bevacizumab (0.016 mg) | Bevacizumab (0.008 mg) | Bevacizumab (0.004 mg) | Bevacizumab (0.002 mg)
Number analyzed (Participants) | 9 | 10 | 16 | 8 | 9 | 5 | 4 | 5
Participants
  Any increase in VEGF | 0 | 0 | 4 | 0 | 2 | 0 | 4 | 1
  Decrease in VEGF by 1% to <25% | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Decrease in VEGF by 25% to <50% | 4 | 2 | 2 | 1 | 1 | 0 | 0 | 1
  Decrease in VEGF by greater than or equal to 50% | 3 | 8 | 9 | 6 | 6 | 5 | 0 | 3

3. Secondary Outcome: Distribution of VEGF Levels
Description: The parents of each infant enrolled in the study will be given the option to participate in a study to measure levels of VEGF and Avastin in the plasma. Participants in this optional study will have blood collected for analysis The distribution of VEGF and Avastin levels (median, range, and quartiles) will be described before injection, and at 2 weeks and 4 weeks post-injection. For each dosage level, at 2, and 4-weeks post-injection, the change from pre-injection will be calculated.
Time Frame: 4 weeks post-injection
Population: In this optional portion of the study, data is available for 61 infants.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab (0.25 mg) | Bevacizumab (0.0125 mg) | Bevacizumab (0.0625 mg) | Bevacizumab (0.031 mg) | Bevacizumab (0.016 mg) | Bevacizumab (0.008 mg) | Bevacizumab (0.004 mg) | Bevacizumab (0.002 mg)
Number analyzed (Participants) | 9 | 10 | 13 | 6 | 8 | 6 | 4 | 5
Participants
  Any increase in VEGF | 1 | 0 | 2 | 1 | 2 | 1 | 4 | 3
  Decrease in VEGF by 1% to <25% | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0
  Decrease in VEGF by 25% to <50% | 3 | 2 | 3 | 1 | 1 | 1 | 0 | 0
  Decrease in VEGF by greater than or equal to 50% | 3 | 7 | 7 | 4 | 4 | 4 | 0 | 2

4. Secondary Outcome: Distribution of Avastin Levels
Description: The parents of each infant enrolled in the study will be given the option to participate in a study to measure levels of VEGF and Avastin in the plasma. Participants in this optional study will have blood collected for analysis The distribution of VEGF and Avastin levels (median, range, and quartiles) will be described before injection, and at 2 weeks and 4 weeks post-injection. For each dosage level, at 2, and 4-weeks post-injection, the change from pre-injection will be calculated, and a 95% confidence interval calculated for the change.
Time Frame: 2 weeks post-injection
Population: Given the optional nature of this blood draw, outcomes were only collected for 56 infants. Given small sample size, we combined all dose levels and reported for those who were enrolled in this optional portion of the study.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Bevacizumab (0.25 mg) | Bevacizumab (0.125 mg) | Bevacizumab (0.0625 mg) | Bevacizumab (0.031 mg) | Bevacizumab (0.016 mg) | Bevacizumab (0.008 mg) | Bevacizumab (0.004 mg) | Bevacizumab (0.002 mg)
Number analyzed (Participants) | 9 | 11 | 19 | 8 | 9 | 0 | 0 | 0
ng/mL | 364 [264 to 424] | 231 [167 to 324] | 292 [111 to 379] | 167 [98 to 274] | 79 [66 to 95] |  |  |

5. Secondary Outcome: Distribution of Avastin Levels
Description: as for outcome 4
Time Frame: 4 weeks post-injection
Population: Given the optional nature of the blood draw and loss to follow up, 4 week data was only collected for 49 infants. Given small sample size, we combined all dose levels and reported for those who were enrolled in this optional portion of the study. Reporting the results overall matches the published MS.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Bevacizumab (0.25 mg) | Bevacizumab (0.125 mg) | Bevacizumab (0.0625 mg) | Bevacizumab (0.031 mg) | Bevacizumab (0.016 mg) | Bevacizumab (0.008 mg) | Bevacizumab (0.004 mg) | Bevacizumab (0.002 mg)
Number analyzed (Participants) | 9 | 11 | 15 | 6 | 8 | 0 | 0 | 0
ng/mL | 281 [242 to 401] | 196 [118 to 258] | 254 [254 to 427] | 115 [81 to 275] | 67 [54 to 99] |  |  |

6. Secondary Outcome: Number of Study Eyes Requiring Additional Treatment/s for ROP
Description: 12-month corrected age calculated as the estimated date of confinement (EDC), or due date, plus 12 months
Time Frame: 12-month corrected age
Population: Eyes, Seven enrolled study eyes and 11 enrolled fellow eyes missing from the table due to lack of 4-week follow-up, including death or deviation. Of these eyes, 5 study eyes and 4 fellow eyes were missing due to death. Eleven additional enrolled fellow eyes missing due to lack of need for initial injection.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab (0.25 mg) | Bevacizumab (0.125 mg) | Bevacizumab (0.0625 mg) | Bevacizumab (0.031 mg) | Bevacizumab (0.016 mg) | Bevacizumab (0.008 mg) | Bevacizumab (0.004 mg) | Bevacizumab (0.002 mg)
Number analyzed (Participants) | 11 | 14 | 24 | 9 | 13 | 9 | 10 | 23
Participants
  Additional Treatment Needed : Severe ROP: Initial Treatment Failure | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 2
  Additional Treatment Needed : Severe ROP: Early Reactivation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Additional Treatment Needed : Severe ROP: Late Reactivation | 2 | 4 | 5 | 0 | 4 | 3 | 3 | 0
  Additional Treatment Needed : Persistent Avascular Retina | 3 | 2 | 3 | 3 | 8 | 2 | 1 | 9
  No Additional Treatment | 6 | 8 | 13 | 6 | 1 | 4 | 5 | 8

7. Secondary Outcome: Any Adverse Events or Complications Since the 4-week Exam
Description: 12-month corrected age calculated as the estimated date of confinement (EDC), or due date, plus 12 months
Time Frame: 12-month corrected age
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab (0.25 mg) | Bevacizumab (0.125 mg) | Bevacizumab (0.0625 mg) | Bevacizumab (0.031 mg) | Bevacizumab (0.016 mg) | Bevacizumab (0.008 mg) | Bevacizumab (0.004 mg) | Bevacizumab (0.002 mg)
Number analyzed (Participants) | 11 | 16 | 24 | 10 | 14 | 9 | 12 | 24
Participants | 4 | 3 | 4 | 1 | 4 | 1 | 5 | 9

8. Secondary Outcome: Visual Fixation Status at 12 Months
Description: 12-month corrected age calculated as the estimated date of confinement (EDC), or due date, plus 12 months
Time Frame: 12-month corrected age
Population: 8 Infants died before exam, exam not completed for 5 participants, and 16 patients were lost to follow up and did not complete.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab (0.25 mg) | Bevacizumab (0.125 mg) | Bevacizumab (0.0625 mg) | Bevacizumab (0.031 mg) | Bevacizumab (0.016 mg) | Bevacizumab (0.008 mg) | Bevacizumab (0.004 mg) | Bevacizumab (0.002 mg)
Number analyzed (Participants) | 10 | 13 | 16 | 6 | 13 | 8 | 10 | 15
Participants
  Central Fixation in Both Eyes | 9 | 13 | 16 | 6 | 11 | 8 | 10 | 12
  Central Fixation in One Eye | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  No Central Fixation in either eye | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 2

9. Secondary Outcome: Proportion of Infants for Whom at Least One Event Was Reported
Description: Adverse events reported at any time during the study will be tabulated for all enrolled infants and coded using the MedRA system. For each dosage level, an estimate and 95% confidence interval of the proportions will be obtained using the exact binomial method
  12-month corrected age calculated as the estimated date of confinement (EDC), or due date, plus 12 months
Time Frame: Enrollment to 12-month corrected age
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab (0.25 mg) | Bevacizumab (0.125 mg) | Bevacizumab (0.0625 mg) | Bevacizumab (0.031 mg) | Bevacizumab (0.016 mg) | Bevacizumab (0.008 mg) | Bevacizumab (0.004 mg) | Bevacizumab (0.002 mg)
Number analyzed (Participants) | 11 | 16 | 24 | 10 | 14 | 9 | 12 | 24
Participants | 6 | 4 | 5 | 1 | 5 | 1 | 5 | 11

10. Secondary Outcome: Proportion of Infants With an Adverse Event Thought by Investigator to be Related to Study Drug
Description: as for outcome 9
Time Frame: Enrollment to 12-month corrected age
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab (0.250 mg) | Bevacizumab (0.125 mg) | Bevacizumab (0.063 mg) | Bevacizumab (0.031 mg) | Bevacizumab (0.016 mg) | Bevacizumab (0.008 mg) | Bevacizumab (0.004 mg) | Bevacizumab (0.002 mg)
Number analyzed (Participants) | 11 | 16 | 24 | 10 | 14 | 9 | 12 | 24
Participants | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0

11. Secondary Outcome: Count of Infants for Whom at Least One Serious Adverse Event Was Reported
Description: Adverse events reported at any time during the study will be tabulated for all enrolled infants and coded using the MedRA system. For each dosage level, an estimate and 95% confidence interval of the proportions will be obtained using the exact binomial method.
Time Frame: Enrollment to 12-month corrected age
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab (0.25 mg) | Bevacizumab (0.125 mg) | Bevacizumab (0.0625 mg) | Bevacizumab (0.031 mg) | Bevacizumab (0.016 mg) | Bevacizumab (0.008 mg) | Bevacizumab (0.004 mg) | Bevacizumab (0.002 mg)
Number analyzed (Participants) | 11 | 16 | 24 | 10 | 14 | 9 | 12 | 24
Participants | 4 | 2 | 3 | 1 | 1 | 0 | 5 | 4

12. Secondary Outcome: Number of Infant Deaths
Description: Adverse events reported at any time during the study will be tabulated for all enrolled infants and coded using the MedRA system.
  12-month corrected age calculated as the estimated date of confinement (EDC), or due date, plus 12 months
Time Frame: Enrollment to 12-month corrected age
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab (0.25 mg) | Bevacizumab (0.125 mg) | Bevacizumab (0.0625 mg) | Bevacizumab (0.031 mg) | Bevacizumab (0.016 mg) | Bevacizumab (0.008 mg) | Bevacizumab (0.004 mg) | Bevacizumab (0.002 mg)
Number analyzed (Participants) | 11 | 16 | 24 | 10 | 14 | 9 | 12 | 24
Participants | 0 | 2 | 2 | 2 | 1 | 0 | 0 | 1

13. Secondary Outcome: Number of Infants With 24-Month Extended Follow Up Exam
Description: A subset of infants enrolled in ROP1 will have extended follow up consisting of one additional office exam with developmental testing.
  This testing will provide a cross-sectional evaluation of visual acuity, refractive error, and development at the adjusted age 24-month visit.
  24-month corrected age calculated as the estimated date of confinement (EDC), or due date, plus 24 months.
Time Frame: 24-month corrected age
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab (0.25 mg) | Bevacizumab (0.125 mg) | Bevacizumab (0.0625 mg) | Bevacizumab (0.031 mg) | Bevacizumab (0.016 mg) | Bevacizumab (0.008 mg) | Bevacizumab (0.004 mg) | Bevacizumab (0.002 mg)
Number analyzed (Participants) | 11 | 16 | 24 | 10 | 14 | 9 | 12 | 24
Participants | 6 | 8 | 15 | 7 | 11 | 6 | 5 | 12

14. Secondary Outcome: Number of Fellow Eyes Requiring Additional Treatment/s for ROP
Description: 12-month corrected age calculated as the estimated date of confinement (EDC), or due date, plus 12 months
Time Frame: 12-month corrected age
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Groups:
- Bevacizumab (0.625 mg); Bevacizumab (0.25 mg); Bevacizumab (0.125 mg); Bevacizumab (0.0625); Bevacizumab (0.031 mg); Bevacizumab (0.016 mg); Bevacizumab (0.008 mg); Bevacizumab (0.004 mg): Dosage of injected Bevacizumab to be studied
Arm/Group | Bevacizumab (0.625 mg) | Bevacizumab (0.25 mg) | Bevacizumab (0.125 mg) | Bevacizumab (0.0625) | Bevacizumab (0.031 mg) | Bevacizumab (0.016 mg) | Bevacizumab (0.008 mg) | Bevacizumab (0.004 mg)
Number analyzed (Participants) | 10 | 14 | 21 | 6 | 10 | 8 | 11 | 18
Participants
  Additional Treatment Needed : Severe ROP: Initial Treatment Failure | 0 | 0 | 3 | 0 | 0 | 1 | 2 | 1
  Additional Treatment Needed : Severe ROP: Early Reactivation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Additional Treatment Needed : Severe ROP: Late Reactivation | 2 | 3 | 5 | 0 | 2 | 2 | 2 | 2
  Additional Treatment Needed : Persistent Avascular Retina | 3 | 3 | 2 | 2 | 7 | 2 | 2 | 8
  No Additional Treatment | 5 | 8 | 11 | 4 | 1 | 3 | 5 | 6

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | Bevacizumab (0.25 mg) | Bevacizumab (0.125 mg) | Bevacizumab (0.0625 mg) | Bevacizumab (0.031 mg) | Bevacizumab (0.016 mg) | Bevacizumab (0.008 mg) | Bevacizumab (0.004 mg) | Bevacizumab (0.002 mg)
All-Cause Mortality (participants affected / at risk) | 0/11 | 3/16 | 2/24 | 2/10 | 1/14 | 0/9 | 0/12 | 1/24
Serious Adverse Events (participants affected / at risk) | 1/11 | 3/16 | 3/24 | 1/10 | 1/14 | 1/9 | 5/12 | 4/24
Other Adverse Events (participants affected / at risk) | 4/11 | 3/16 | 4/24 | 1/10 | 4/14 | 1/9 | 5/12 | 9/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (0.25 mg) (N=11) | Bevacizumab (0.125 mg) (N=16) | Bevacizumab (0.0625 mg) (N=24) | Bevacizumab (0.031 mg) (N=10) | Bevacizumab (0.016 mg) (N=14) | Bevacizumab (0.008 mg) (N=9) | Bevacizumab (0.004 mg) (N=12) | Bevacizumab (0.002 mg) (N=24)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Apnoea Neonatal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Potassium increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic Respiratory Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Feeding Intolerance (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal tube insertion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrostomy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic Failure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infantile apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Penumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Hypertension (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyloric stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 2 (3)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Retinal Detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal neovascularisation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small Intestine Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tricuspid valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (0.25 mg) (N=11) | Bevacizumab (0.125 mg) (N=16) | Bevacizumab (0.0625 mg) (N=24) | Bevacizumab (0.031 mg) (N=10) | Bevacizumab (0.016 mg) (N=14) | Bevacizumab (0.008 mg) (N=9) | Bevacizumab (0.004 mg) (N=12) | Bevacizumab (0.002 mg) (N=24)
Any Adverse Event (Eye disorders) | 4 | 3 | 4 | 1 | 4 | 1 | 5 | 9 — An adverse event is any untoward medical occurrence in a study participant, irrespective of whether or not the event is considered treatment-related.
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Apnoea neonatal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterameia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Candida infection (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract cortical (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract operation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clonus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Congenital coronary artery malformation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corneal Disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Feeding Intolerance (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal Skin Infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal tube insertion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemangioma of Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hernia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydrocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iris Adhesions (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacrimation Increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngomalacia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic Alkalosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal Detachment (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Retinal Disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal Haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 1 (1)
Retinal Vein Occlusion (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal Burn (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT02390531/Prot_001.pdf
  • Statistical Analysis Plan (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT02390531/SAP_002.pdf
  • Informed Consent Form (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/31/NCT02390531/ICF_000.pdf